CLINICAL TRIAL: NCT02991898
Title: Adoptive Transfer of T Regulatory Cell for Suppression of Acute Graft-vs-Host-Disease After an Umbilical Cord Blood Transplant for Hematologic Malignancies
Brief Title: Adoptive TReg Cell for Suppression of aGVHD After UCB HSCT for Heme Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Considering new technology for product.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016LS107; MT2016-17 (Other: University of Minnesota Blood and Marrow Transplant Program)
Record Dates: First submitted 2016-12-07; First posted 2016-12-14 (Estimated); Results first posted 2020-07-24 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Acute Lymphoblastic Leukemia; Burkitt Lymphoma; Natural Killer Cell Malignancies; Chronic Myelogenous Leukemia; Myelodysplastic Syndromes; Large-cell Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Marginal Zone B-Cell Lymphoma; Follicular Lymphoma; Lymphoplasmacytic Lymphoma; Mantle-Cell Lymphoma; Prolymphocytic Leukemia; Hodgkin Lymphoma; Multiple Myeloma; Acute Myelogenous Leukemia; Biphenotypic Leukemia; Undifferentiated Leukemia
Keywords: CML; MDS; CLL; ALL; AML
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Dendritic Cell Sarcoma, Interdigitating; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Prolymphocytic; Hodgkin Disease; Multiple Myeloma; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treg Infusion (Experimental): The Treg cell infusion is given no sooner than 1 hour, but within 24 hours after the 2nd cord blood infusion
  Interventions: Biological: Infusion of Treg

INTERVENTIONS:
Biological: Infusion of Treg — Allopurinol on day -7 to day 0 Cyclophosphamide 50 mg/kg IV over 2 hours on day -6 Fludarabine 30mg/m2 IV over 1 hour on day -6, -5, -4, -3, and -2 Total Body Irradiation 200 cGy as a single dose
  Sirolimus 8mg-12mg oral loading dose followed by single dose 4mg/day. Levels are to be monitored 3 times/week in the first week, weekly until day +60, and as clinically indicated until day +100 post-transplantation.
  Mycophenolate Mofetil (MMF) 3 gram/day IV/PO divided in 2 or 3 doses. Stop MMF at day +30 or 7 days after neutrophil recovery, whichever day is later, if no acute GVHD.
  DUCBT followed Tregs - double umbilical cord blood transplant (FIRST) followed by the Treg cell infusion (SECOND) no sooner than 1 hour, but within 24 hours after the 2nd cord blood infusion.
  Other Names: T regulatory cells

SUMMARY:
This is a single center pilot study of a non-myeloablative umbilical cord blood transplant for the treatment of a hematological malignancy with a single infusion of T regulatory (Treg) given shortly after UCB transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥18, but < 70 years of age with no matched 7/8 or 8/8 sibling donor - patients ≥ 70 and ≤ 75 years of age may be eligible if they have a Co-Morbidity score ≤ 2 (http://www.qxmd.com/calculate-online/hematology/hct-ci)
* UCB unit(s) composing the graft will be selected according to the current University of Minnesota umbilical cord blood graft selection algorithm and an additional cord blood unit to be used as the source to manufacture the Treg product. This UCB unit must be matched at 4-6/6 to the patient, considering HLA-A, B at the antigen level and DRB1 at the allele level
* Acute Leukemias: Must be in remission by morphology. Also a small percentage of blasts that is equivocal between marrow regeneration versus early relapse are acceptable provided there are no associated cytogenetic markers consistent with relapse. Refer to Section 5.2 for complete definitions.
* Burkitt's Lymphoma in CR2 or subsequent CR
* Natural Killer Cell Malignancies
* Chronic Myelogenous Leukemia: all types except refractory blast crisis. Chronic phase patients must have failed at least two different tyrosine-kinase inhibitors (TKIs), or been intolerant to all available TKIs or have T315I mutation.
* Myelodysplastic Syndrome: IPSS INT-2 or High Risk; R-IPSS High or Very High; WHO classification: RAEB-1, RAEB-2; Severe Cytopenias: ANC < 0.8, Anemia or thrombocytopenia requiring transfusion; Poor or very poor risk cytogenetics based on IPSS or R-IPSS definitions; therapy-related MDS. Blasts must be be < 5%, preferably < 20% blasts by morphology by bone marrow aspirate morphology.. If ≥ 5% blasts, chemotherapy for cytoreduction to <5% blasts prior to transplantation may be considered.
* Chronic myeloid neoplasms, including but not limited to CMML with blasts must around 5% blasts, preferably < 20% blasts by morphology by bone marrow aspirate morphology. If ≥5% blasts, chemotherapy for cytoreduction to <5% blasts prior to transplantation may be considered.
* Large-Cell Lymphoma, Hodgkin Lymphoma and Multiple Myeloma with chemotherapy sensitive disease that has failed or patients who are ineligible for an autologous transplant.
* Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL), Marginal Zone B-Cell Lymphoma, Follicular Lymphoma, which have progressed within 12 months of achieving a partial or complete remission. Patients who had remissions lasting > 12 months are eligible after at least two prior therapies. Patients with bulky disease should be considered for debulking chemotherapy before transplant. Patients with refractory disease are eligible, unless has bulky disease and an estimated tumor doubling time of less than one month.
* Lymphoplasmacytic Lymphoma, Mantle-Cell Lymphoma, Prolymphocytic Leukemia are eligible after initial therapy if chemotherapy sensitive.
* Patients must have undergone an autologous transplant ≤ 12 months prior to transplant on this study or have received multi-agent or immunosuppressive chemotherapy within 3 months of the preparative regimen.

Performance Status, Organ Function, Contraception Use

* Karnofsky score ≥ 70% (Appendix II)
* Adequate organ function within 14 days (30 days for cardiac and pulmonary) of registration on-study defined as:

  * Renal: creatinine ≤ 2.0 mg/dL, for patient with a creatinine > 1.2 mg/dL or a history of renal dysfunction an estimated glomerular filtration rate ≥ 40 mL/min/1.73 m2 is required
  * ALT, AST and alkaline phosphatase ≤ 5 x upper limit of normal and total bilirubin ≤ 2.5 mg/dL except for patients with Gilbert's syndrome or hemolysis
  * Pulmonary function: DLCO, FEV1, FVC ≥ 40% predicted, and absence of O2 requirements.
  * Cardiac: Absence of decompensated congestive heart failure, or uncontrolled arrhythmia and left ventricular ejection fraction ≥ 40%.
* Sexually active females of childbearing potential and males with partners of child-bearing potential must agree to use adequate birth control during study treatment.
* Voluntary written consent

Exclusion Criteria:

* Untreated active infection
* History of HIV infection
* Pregnant or breast feeding. The agents used in this study may be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. Females of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy
* Prior allogeneic transplantation
* Less than 3 months from myeloablative conditioning for autologous transplantation (if applicable)
* Evidence of progressive disease by imaging modalities or biopsy - persistent PET activity, though possibly related to lymphoma, is not an exclusion criterion in the absence of CT changes indicating progression.
* CML in blast crisis
* Large cell lymphoma, mantle cell lymphoma and Hodgkin disease that is progressing on salvage therapy.
* Active central nervous system malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Brunstein, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treg Infusion
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treg Infusion
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Survived
Description: Count of patients who survived 2 years post intervention
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treg Infusion
Number analyzed (Participants) | 3
Participants | 1

2. Secondary Outcome: Number of Participants With Grade II-IV aGVHD
Description: Probability of grade II-IV aGVHD
Time Frame: Assessed weekly until day 100, then day 180, 360
Measure: Count of Participants; unit: Participants
Arm/Group | Treg Infusion
Number analyzed (Participants) | 3
Participants | 2

3. Secondary Outcome: Number of Participants Experiencing Treatment Related Mortality (TRM)
Description: Evaluated with descriptive statistics and plots or cumulative incidence curves if enough evaluable patients are available for time-to-event endpoints.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treg Infusion
Number analyzed (Participants) | 3
Participants | 0

4. Secondary Outcome: Number of Participants Who Experienced Relapse
Description: as for outcome 3
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treg Infusion
Number analyzed (Participants) | 3
Participants | 1

5. Secondary Outcome: Number of Participants With Incidence of Bacterial, Viral and Fungal Infections
Description: as for outcome 3
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treg Infusion
Number analyzed (Participants) | 3
Participants
  Bacterial | 1
  Viral | 2
  Fungal | 0

6. Secondary Outcome: Number of Participant With Detectable Treg Cells at d14
Description: The proportion of patients with detectable Treg cells at day 14 post infusion
Time Frame: 14 days
Population: Samples were not analyzed, and so data not available for reporting.
Arm/Group | Treg Infusion
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Immune Reconstitution
Description: The proportion of patients with immune reconstitution. Continuous endpoints will be described by medians, ranges and interquartile ranges as well as means and standard deviations if normally distributed.
Time Frame: Assessed at Day 4, weekly for 8 weeks
Population: Samples were not analyzed, and so data not available for reporting.
Arm/Group | Treg Infusion
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants Experiencing Treg Cell Infusion Toxicity
Description: Incidence of Adverse Events
Time Frame: 48 hours post infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Treg Infusion
Number analyzed (Participants) | 3
Participants | 2

9. Secondary Outcome: Length of Treg Survival
Description: Length of Treg survival after infusion of Treg.
Time Frame: 24 hours post infusion
Population: Samples were not analyzed, and so data not available for reporting.
Arm/Group | Treg Infusion
Number analyzed (Participants) | 0

10. Secondary Outcome: Percentage of Donor Cell Chimerism
Description: The incidence of chimerism in patients treated
Time Frame: Day +100
Measure: Mean (Full Range); unit: percentage of donor cells
Arm/Group | Treg Infusion
Number analyzed (Participants) | 3
percentage of donor cells | 72 [50 to 100]

11. Secondary Outcome: Number of Participants Survived One Year Post-transplant
Description: The probability of survival, one year post-treatment
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treg Infusion
Number analyzed (Participants) | 3
Participants | 2

12. Secondary Outcome: Number of Participants With Neutrophil Recovery
Description: The incidence of neutrophil recovery, that is return of neutrophil counts to ≥ 5 X 10^8/L in treated patients
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Treg Infusion
Number analyzed (Participants) | 3
Participants | 2

13. Secondary Outcome: Number of Participants With Platelet Recovery
Description: The incidence of platelet recovery (return of platelet counts to > 20,000/μL) in treated patients
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treg Infusion
Number analyzed (Participants) | 3
Participants | 2

14. Secondary Outcome: Number of Participants With Chronic GVHD
Description: The incidence of chronic GVHD in treated patients after one year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treg Infusion
Number analyzed (Participants) | 3
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Treg Infusion
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treg Infusion (N=3)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Cytokine release syndrome (Vascular disorders) | 1 (1)
Graft Versus Host Disease (Immune system disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treg Infusion (N=3)
Hypertension (Cardiac disorders) | 1 (7)
Chills (General disorders) | 1 (2)
Edema Limbs (General disorders) | 1 (4)
Fatigue (General disorders) | 1 (2)
Febrile neutropenia (General disorders) | 1 (3)
Fever (General disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT02991898/Prot_SAP_000.pdf